CLINICAL TRIAL: NCT07239869
Title: An AI Robot-assisted Tailored Activity Programme for Improving the Physical Inactivity of People With Dementia and Their Informal Caregivers
Brief Title: A Robot-assisted Tailored Activity Programme for People With Dementia and Their Caregivers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P0044775
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Dementia; Caregiver; Physical Activity; Psychological Well Being
MeSH Terms: conditions — Dementia; Motor Activity; Psychological Well-Being | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Tweleve weeks of robot-assisted tailored activity programme
  Interventions: Other: Intervention
- Control (Other): Usual care provided by community centers
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — 12 weeks of robot assisted tailored activity programme
  Arms: Intervention
Other: Control — Usual care provided by community centers
  Arms: Control

SUMMARY:
To assess the feasibility and preliminary efficacy of the tailored activity programme on improving the physical inactivity of the caregiving dyads.

DETAILED DESCRIPTION:
This is a two-arm pilot randomized controlled trial evaluating the feasiblity and preliminary efficacy of the robot-assisted tailored activity programme on improving the physical inactivity of people with dementia and their caregivers. Sixty dyads will be rectuited. Participants in the intervention group will receive a 12-week tailored activity programme, while those in the control group will receive usal community care services. Outcomes including feasibility of the tailored acitivity programme, physical activity levels, self-efficacy in physical activity, dyadic quality of life, neuropsychiatric somptoms, and psychological wellbeing will be measured at baseline and immediately post intervention.

ELIGIBILITY:
Inclusion Criteria for people with dementia:

* mild to moderate stage dementia at a standardized mini-mental state examination score (MMSE) higher than 10;
* be able to walk independently;
* being physically inactive (categorized as "low/inactive" by the International Physical Activity Questionnaire);
* free from other medical/functional conditions that would limit physical activity.

Exclusion Criteria for people with dementia:

* high risk of falling (Berg Balance Scale <45);
* not be suitable for doing physical activity as recommended by the primary care physician;
* currently involved in another interventional study involving physical exercise;
* had acute hospitalization >3 times in the past year.

Inclusion Criteria for caregivers:

* primary informal caregivers who reside with the of the person with dementia;
* have provided care for more than six months;
* have no intention to send the care recipient to nursing homes in the next six months;
* being physically inactive;
* use a smartphone.

Exclusion Criteria for caregivers:

* caregivers with unstable physical or mental conditions;
* cannot communicate logically;
* not suitable for doing physical activity as recommended by a primary care physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in physical activity | Pre-intervention and immediately post-intervention
  Physical activity will be measured with the Chinese version of the International Physical Activity Questionnaire short version (IPAQ-C, short). The IPAQ-C is a 9-item instrument with good reliability and validity. Objective mesures will include number of steps, movement distance, sedentary minutes, inactive minutes collected with an activity tracker.

SECONDARY OUTCOMES:
Changes in self-efficacy in physical activity | Pre-intervention and immediately post-intervention
  Self-efficacy in physical activity will be measured with a Likert 6-point scale covering three different types of self-efficacy. This instrument demonstrated satisfactory internal consistency. Higher scores indicate higher self-efficacy in physical activity.
Changes in quality of life | Pre-intervention and immediately post-intervention
  Dyadic quality of life will be measured with the 12-item Short Form Survey (SF-12). Higher scores indicate better quality of life
Changes in neuropsychiatric symptoms of people with dementia | Pre-intervention and immediately post-intervention
  People with dementia's neuropsychiatric symptoms will be measured with the Neuropsychiatric Inventory (NPI). NPI evaluates 12 common neuropsychiatric disturbances in dementia. The Chinese version was reliable. Higher scores indicate worse symptoms
Changes in psychological well-being | Pre-intervention and immediately post-intervention
  Dyads' psychological well-being will be measured with the Depression Anxiety Stress Scale-21 (DASS-21). DASS-21 includes 3 subscales (stress, anxiety, and depression), and has demonstrated good reliability among the Chinese population. Higher scores indicate poorer psychological wellbeing and more psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No